CLINICAL TRIAL: NCT01538706
Title: Hospital-based Home Care for Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Helena Hansson, Clinial Researcher and Nurse Specialist, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 959584438
Record Dates: First submitted 2011-11-09; First posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Neoplasms; Children
Keywords: Hospital-based home care; Pediatric oncology
MeSH Terms: conditions — Neoplasms | interventions — Home Care Services, Hospital-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hospital-based home care (Experimental): Patients were included if below the age of 18, had been diagnosed with any type of cancer at least one month prior to inclusion, on intravenous anticancer therapy with a curative intent, and the parent was fluent in speaking and reading Danish. Patients living within a radius of 50 kilometres from the hospital were assigned to the home care program. Moreover, patients were assigned to one of three groups according to the geographical distance from the hospital and timing of the inclusion period: (1) home care group if participating in the program, (2) historical standard care group for an eight-month period before the program started regardless of their residence distance from the hospital, and (3) concurrent standard care group if living more than 50 km from the university hospital.
  Interventions: Other: Hospital-based home care

INTERVENTIONS:
Other: Hospital-based home care — Low-intensive intravenous antibiotics b) intravenous low-toxic chemotherapy c) blood samples drawn from the central venous catheter or peripheral vein d) subcutaneous injections e) nutrition treatment f) pain management (e.g. controlling an intravenous morphine pump g) supportive care e.g. changing dressings.

SUMMARY:
The purpose of this non-randomized controlled intervention study was to evaluate the effects of a hospital-based home care program for children with cancer at a university hospital in Denmark. The hypothesis was that hospital-based home care could replace an out-patient visit or an in-patient admission without increasing the incidence of adverse events and costs. Furthermore, to enhance the children's quality of life and the psychosocial impact on the family.

DETAILED DESCRIPTION:
Hospital-based home care for children with cancer is widely used but controlled studies are relatively rare and the evidence base is limited. This prospective non-randomized controlled intervention study aimed to evaluate hospital-based home care for children with cancer.

A hospital-based home care program was conducted August 2008 - December 2009. Participants were children with cancer and their parents. The intervention group received part of their therapy, such as intravenous chemotherapy and antibiotics, as home care by a hospital-based home care nurse with paediatric-oncology experience. Children in the control group received all their treatment at the hospital.

Fifty-one children between 0 and 18 years were included in the home care program, and 47 children were included in the control group. After each home visit the parents answered a questionnaire. The results from 657 questionnaires showed that 100% were very satisfied or satisfied with home care and all would choose home care again, if offered as an option. There were no deaths or adverse effects of intravenous chemotherapy or antibiotics. A cost analysis based on the expenses associated with home care in correlation with standard cost of inpatient admissions and outpatient visits showed that the hospital-based home care programme was economically equal. The children's and the families' quality of life may be enhanced. The results indicate that the hospital-based home care program is safe, economically neutral and the parents' satisfaction with the program is major.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cancer
* First-line treatment with intravenous therapy with a curative intent
* Have not received a haematopoietic stem cell transplantation
* Child and parent(s) speak and read Danish

Exclusion Criteria:

* End-of-life treatment
* Critical medical condition

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 17 months
  At each home visit, the hospital-based home care nurse recorded details on the HBHC visits and safety according to the mandatory hospital guidelines for registrations of adverse events such as acute deteriorations of the general condition, and any medical errors.

SECONDARY OUTCOMES:
Costs of the intervention | 17 months
  The costs for the health care service were evaluated by comparing the hospital-based home care related operational e.g. petrol and pay roll costs plus overhead costs, with the billed costs for an out-patient visit or in-patient admission at the hospital.
Healthrelated quality of life of the child with cancer | At inclusion and 3 months after
  A questionnaire booklet was developed to compare the psychosocial impact on the child and the family with home care and standard care. The child's general health-related quality of life was assessed by the PedsQL 4.0 Generic Core Scale, which consists of four dimensions and a total score of all dimensions is computed as well as a physical and psychosocial summary score. The child's disease-specific health-related quality of life was assessed by the PedsQL 3.0 Cancer Module, which consists of seven dimensions without a total score.
Psychosocial impact of the family with a child of cancer | At inclusion and 3 months after
  A questionnaire booklet was developed to compare the psychosocial impact on the child and the family with home care and standard care. The psychosocial impact on the family was assessed by PedsQL 2.0 Family Impact Module, which consists of 8 dimensions with a total score as well as the parent's health-related quality of life and family functioning summary score.
Participants' satisfaction with health care | At inclusion and 3 months after
  A questionnaire booklet was developed to compare the psychosocial impact on the child and the family with home care and standard care. The participants' satisfaction with health care was assessed by PedsQL Healthcare Satisfaction Generic Module measures the parents'/guardians' satisfaction with health care in general in six dimensions: information, inclusion of family, communication, technical skills, emotional needs, and overall satisfaction. A total score of all dimensions is computed.
Participants' satisfaction with the hospital-based home care program | 12 months
  A one-page evaluation form to measure the parents' and children's perceptions of security, satisfaction with home care and preference for care was developed with a 5-point Likert- scale ranging from not at all to very much. The parents' also scored overall preference for standard vs. home care was scored with two alternative responses (yes or no) and they were asked whether they would choose a home care visit again instead of a corresponding hospital visit if they had the opportunity.
  The evaluation forms were collected after each home visit only during the first 12 months of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Hansson, MSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen university hospital, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Result] Hansson H, Kjaergaard H, Schmiegelow K, Hallstrom I. Hospital-based home care for children with cancer: a qualitative exploration of family members' experiences in Denmark. Eur J Cancer Care (Engl). 2012 Jan;21(1):59-66. doi: 10.1111/j.1365-2354.2011.01280.x. Epub 2011 Aug 18. PMID 21848580